CLINICAL TRIAL: NCT05651516
Title: Effects of Opioid Use Disorder and Non-fatal Overdose on Tau Pathology; a [18F]PI-2620 PET/CT Study
Brief Title: Tau PET Imaging in Opioid Use Disorder
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 852095
Record Dates: First submitted 2022-12-01; First posted 2022-12-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Opioid-Related Disorders
Keywords: Tau; PET/CT
MeSH Terms: conditions — Opioid-Related Disorders; Pick Disease of the Brain | interventions — PI-2620

STUDY DESIGN:
Intervention Model Description: The analyses for the three aims will use analysis of variance to test for group differences among the three groups (OUD/OD+, OUD/OD-, HC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tau PET/CT (Experimental): PET/CT imaging will be used to evaluate the uptake of tau in the brain using the investigational radiotracer [18F]PI-2620. Each subject will have one [18F]PI-2620 positron emission tomography/computed tomography (PET/CT) scan performed.
  Participants will undergo approximately 30 minutes of static PET scanning of the brain and body starting approximately 45 minutes post injection of [18F]PI-2620. All images will be corrected for scatter and measured photon attenuation and reconstructed using standard reconstruction techniques. Standardized uptake value ratio (SUVr), the ratio of regional to reference uptake, will be calculated with cerebellum as reference, where NFTs are generally not present in neurodegenerative disorders, hence likely not in OUD.
  Subjects in all three groups undergo a brain MRI including a structural MRI functional reactivity to an episodic memory task, and undergo a comprehensive neurocognitive battery.
  Interventions: Drug: 18F-PI-2620 PET/CT

INTERVENTIONS:
Drug: 18F-PI-2620 PET/CT — PET/CT imaging will be used to evaluate the uptake of tau in the brain using the investigational radiotracer [18F]PI-2620. Each subject will have one [18F]PI-2620 positron emission tomography/computed tomography (PET/CT) scan performed.
  Other Names: PI-2620

SUMMARY:
The investigators plan to enroll up to 60 adult subjects in this study. There will be three groups of up to 20 subjects each in this study.

Group 1: individuals with OUD and a history of at least one opioid-related OD in the past 5 years that required naloxone treatment reversal: OUD/OD+ Group 2: individuals with OUD without a lifetime history of opioid-related OD OUD/OD- Group 3: Healthy controls without a lifetime OUD: HCs PET/CT imaging will be used to evaluate the uptake of tau in the brain using the investigational radiotracer [18F]PI-2620. Each subject will have one [18F]PI-2620 positron emission tomography/computed tomography (PET/CT) scan performed.

DETAILED DESCRIPTION:
Participants will undergo approximately 30 minutes of static PET scanning of the brain and body starting approximately 45 minutes post injection of [18F]PI-2620. All images will be corrected for scatter and measured photon attenuation and reconstructed using standard reconstruction techniques. Standardized uptake value ratio (SUVr), the ratio of regional to reference uptake, will be calculated with cerebellum as reference, where NFTs are generally not present in neurodegenerative disorders, hence likely not in OUD.

Subjects in all three groups undergo a brain MRI including a structural MRI functional reactivity to an episodic memory task, and undergo a comprehensive neurocognitive battery.

The investigators will draw up to 60 mL of venous blood prior to injection that will be used to measure peripheral blood markers of phosphorylated tau, inflammation, and ApoE genotyping. The results of these research tests will not be given to the subject, will not be included in the medical record and will not be used in the subject's clinical management.

Additional measures will be collected: measures of substance use and related behaviors, psychological and subjective measures, neurocognitive measures and OUD-related health outcomes for correlation with the imaging results.

ELIGIBILITY:
Inclusion Criteria:

OUD OD- group:

1. 18-60 years-old
2. Informed of the investigational nature of this study and able to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
3. Participants meet for lifetime OUD and are currently in medication-assisted treatment for OUD, which must include being on a stable dose of medication for at least 30 days prior to the screening visit.
4. No lifetime history of OD per self-report, Drug Overdose Questionnaire, and/or medical record review.

OUD OD+ group:

1. 18-60 years-old
2. Informed of the investigational nature of this study and able to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
3. Participants meet for lifetime OUD and are currently in medication-assisted treatment for OUD, which must include being on a stable dose of medication for at least 30 days prior to the screening visit.
4. A history of at least 1 opioid OD that required naloxone reversal that occurred up to 5 years prior to study enrollment, as per self-report, Drug Overdose Questionnaire, and/or medical record review.

Healthy Control (HC) group:

1. 18-60 years-old
2. Informed of the investigational nature of this study and able to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
3. Must have never met lifetime history for Alcohol Use Disorder, Substance Use Disorder --other than cannabis, tobacco or nicotine use disorder (as per DSM-5) and not used an opioid for any reason in the 30 days prior to screening by self-report, medical record review, and urine drug testing at screening.
4. Must provide a negative urine drug screen on the day of the screening, MRI and PET scan visits for all substances (other than cannabis).

Exclusion Criteria:

1. HIV infection confirmed by an on-site rapid HIV test at screening. HIV affect neurocognitive function, even in otherwise asymptomatic individuals, which can confound the results of MRI testing.
2. The urine drug screening & pregnancy test (for women of child-bearing potential) at the screening visit, MRI visit, and PET/CT scan visits must be negative for pregnancy (all groups) or will be deemed ineligible to participate. Participants in the healthy control group with a positive drug screen will be ineligible.
3. At screening, the participant's weight is >350 lb.
4. Self-reported claustrophobia, which in the opinion of an investigator would interfere with acquisition of the structural MRI required for PET co-registration, and/or the PET scan itself.
5. Contraindications to MRI (e.g., metal in the body that cannot be removed and is not MRI compatible). An MRI screening form will be completed during screening to identify contraindications.
6. Screening lab values that indicate significant organ dysfunction that in the opinion of an investigator could compromise participant safety or successful participation in the study.
7. History of epilepsy or seizure disorder (that are not a result of substance use or substance withdrawal in OUD+ groups) as assessed by medical record review or self-report.
8. History of head trauma that in the opinion of an investigator may interfere with the uptake of applicable radiotracer as assessed by medical record review or self-report.
9. Current serious psychiatric disorder (bipolar disorder, schizophrenia, psychotic disorder, eating disorder, or major depressive disorder with suicidal ideation or psychotic features) identified by medical record review, clinical examination or structured psychiatric interview that could interfere with study participation or make it hazardous for the participant or staff to perform study procedures.
10. Self-reported heavy daily use of psychoactive substances in the past 30 days (prior to the screening visit), such as stimulants, cocaine, but not including nicotine, caffeine, cannabis (or opioids in the OUD groups) that could interfere with study performance.
11. Not able to provide a breath alcohol level of 0.000 (tested with handheld breath analyzer) at the screening, MRI and/or PET scan visits.
12. Inability to tolerate imaging procedures as determined by an investigator or treating physician
13. Any current medical condition, illness, or disorder assessed by medical record review and/or self-report that is considered by a physician or investigator to potentially compromise participant safety or their successful participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value ratio (SUVr), | 8 weeks
  • [18F]PI-2620PET SUVr regional uptake (occipital cortex, medial parietal/posterior cingulate cortex, temporoparietal cortex, medial temporal lobe, frontal lobes).

SECONDARY OUTCOMES:
MRI cortical volume | 8 weeks
  MRI cortical volume
MRI cortical thickness | 8 weeks
  MRI cortical thickness

OTHER OUTCOMES:
Neurocognitive test results | 8 weeks
  To determine the effects of OUD and non-fatal opioid OD on episodic memory performance. While in the MRI scanner, all participants will undergo a hippocampus-dependent visual episodic memory task during a functional MRI scan, for which hippocampal BOLD responses correlate with entorhinal [18F]PI-2620 binding in Alzheimer's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Nasrallah, MD, PhD, Principal Investigator — Univeristy of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No